CLINICAL TRIAL: NCT00766142
Title: Clinical Phase II Study Evaluating Systemic Chemotherapy in Combination With Cetuximab as Adjuvant Treatment in Patients With Completely Surgically Resected Peritoneal Carcinomatosis of Colorectal Origin
Brief Title: Chemotherapy and Cetuximab in Patients Undergoing Surgery for Peritoneal Carcinomatosis From Colorectal Cancer
Acronym: COCHISE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In 2008, new data highlighted that Cetuximab had no efficacy in case of KRAS mutation. As such, eligibility criteria were revised and limited to KRAS wild-type. Inclusions were thus slown down considerably, and the trial was stopped.
Sponsor: Institut Bergonié (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Centre Alexis Vautrin, Nancy (Other); Centre Leon Berard (Other); Institut Cancerologie de l'Ouest (Other); Hôpital Haut-Lévêque (Other); Clinique Médicale de Francheville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB-2007-20; IB-COCHISE-I (Other: Institut Bergonié); EUDRACT-2006-003900 (Registry Identifier: EUDRACT); MERCK-IB-COCHISE-I (Other: MERCK)
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer; Primary Peritoneal Cavity Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage IV rectal cancer; peritoneal carcinomatosis
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Peritoneal Neoplasms | interventions — Cetuximab; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: Combination Chemotherapy and Cetuximab in Treating Patients Undergoing Surgery for Peritoneal Carcinomatosis From Colorectal Cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + Cetuximab (Experimental): Surgery + Chemotherapy + Cetuximab
  Interventions: Biological: cetuximab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: adjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Biological: cetuximab
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving more than one drug (combination chemotherapy) together with cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well chemotherapy given together with cetuximab works in treating patients undergoing surgery to remove peritoneal carcinomatosis from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of systemic chemotherapy and cetuximab, in terms of progression-free survival at 3 years, in patients with completely resected peritoneal carcinomatosis of colorectal origin.

Secondary

* Determine the therapeutic strategy among patients who are or are not fit to receive chemotherapy.
* Determine progression-free survival at 5 years and overall survival at 3 and 5 years in these patients.
* Determine the overall tolerability (mortality, morbidity) of this regimen, including surgery, in these patients.

OUTLINE: This is a multicenter study.

Patients undergo complete resection of the peritoneal carcinomatosis. Beginning 4-8 weeks after surgery, patients receive cetuximab IV over 2.5 hours. Patients also receive FOLFOX chemotherapy comprising oxaliplatin IV and leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46 hours. Treatment repeats every 2 weeks for up to 12 courses.

After completion of study therapy, patients are followed every 4 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma meeting the following criteria:

  * Exclusively peritoneal carcinomatosis (no other metastases)
  * Resectable disease
* Primary tumor may be same in the same location as another synchronous carcinomatosis
* Patients with metastatic disease who have been in complete remission for more than 1 year are eligible regardless of prior chemotherapy

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 10 g/dL
* Bilirubin ≤ 1.25 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Creatinine ≤ 1.25 times ULN
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No allergy, hypersensitivity, or other contraindication to leucovorin calcium, oxaliplatin, or fluorouracil
* No other noncancerous disease that would preclude study therapy
* Good nutritional status
* No sensitive peripheral neuropathy with functional impairment
* No hypoplasia or bone marrow failure
* No clinically significant cardiovascular disease within the past year (e.g., unstable angina or myocardial infarction)
* No other cancer within the past 5 years unless in complete remission with the exception of cervical carcinoma in situ or basal cell cancer
* No patients deprived of liberty or under supervision
* No psychological, social, familial, or geographical reasons prohibiting follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 1 year since prior adjuvant chemotherapy, including prior therapy with oxaliplatin and/or cetuximab
* No prophylactic phenytoin (Dihydan®, Dilantin®)
* No prior yellow fever vaccine
* More than 1 month since participation in another study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05-01; Primary Completion 2013-09-17 (Actual); Study Completion 2013-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Evrard, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Evrard S, Desolneux G, Bellera C, Esnaud T, Becouarn Y, Collet D, Chafai N, Marchal F, Cany L, Lermite E, Rivoire M, Mathoulin-Pelissier S. Systemic chemotherapy plus cetuximab after complete surgery in the treatment of isolated colorectal peritoneal carcinoma: COCHISE phase II clinical trial. BMC Res Notes. 2019 Jul 22;12(1):450. doi: 10.1186/s13104-019-4476-9. PMID 31331370

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy + Cetuximab: * Cetuximab 500 mg/m² IV
  * Oxaliplatine 85 mg/m² IV
  * L-folinique Acid 200 mg/m² (or 400 mg/m² for DL) IV
  * 5-FU bolus 400 mg/m² IV
  * 5-FU continu 2400 mg/m² IV. One cycle = 14 days. Up to 12 cycles.
Period: Overall Study
Arm/Group | Chemotherapy + Cetuximab
Started | 18
Completed | 14
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Population: Population with resection after surgery
Arm/Group | Chemotherapy + Cetuximab
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 14

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS) Time
Description: Progression-free survival time is defined as the time from the date of surgery to the date of progression (as per RECIST v1.1) or death of any cause, whichever occurs first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Since surgery, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy + Cetuximab
Number analyzed (Participants) | 14
months | 12.2 [6.5 to 17.3]

2. Secondary Outcome: 30-day Mortality Rate
Description: Rate of deaths observed within 30 days of surgery
Time Frame: from the date of surgery up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Cetuximab
Number analyzed (Participants) | 14
Participants | 0

3. Secondary Outcome: Mean Number of Adverse Events Per Patient, Within 30 Days of Surgery
Time Frame: from the date of surgery up to 30 days
Measure: Mean (95% Confidence Interval); unit: adverse events
Arm/Group | Chemotherapy + Cetuximab
Number analyzed (Participants) | 14
adverse events | 0.93 [0 to 3.7]

4. Secondary Outcome: Overall Survival (OS) Time
Description: OS is the delay between surgery and death
Time Frame: from surgery, up to five years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy + Cetuximab
Number analyzed (Participants) | 14
months | 41.5 [18.4 to 60]

ADVERSE EVENTS:
Time Frame: from surgery, up to 5 years
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term,
Groups:
- Chemotherapy + Cetuximab: cetuximab
  fluorouracil
  leucovorin calcium
  oxaliplatin
  adjuvant therapy
  therapeutic conventional surgery
Arm/Group | Chemotherapy + Cetuximab
All-Cause Mortality (participants affected / at risk) | 8/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy + Cetuximab (N=14)
Vascular disorders - Other (Vascular disorders) | 1 (1) — Vascular disorders - Other
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Urinary fistula (Renal and urinary disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy + Cetuximab (N=14)
Allergic reaction (Immune system disorders) | 2 (2)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
White blood cell decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Fatigue (General disorders) | 10 (10)
Fever (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Weight loss (Investigations) | 1 (1)
burn (Injury, poisoning and procedural complications) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Flushing (Vascular disorders) | 4 (4)
Injection site reaction (General disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 9 (10)
Small intestinal mucositis (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (3)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (16)
Pain (General disorders) | 2 (2)
Pain, other (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes